CLINICAL TRIAL: NCT05873530
Title: Circadian Modulation of Grape Consumption and Oxidative Stress Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Idaho State University (Other)
Responsible Party: Principal Investigator, Cynthia Blanton, Professor, Idaho State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB-FY2021-264
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Oxidative Stress
MeSH Terms: interventions — whole grape extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time (Experimental): Morning or evening
  Interventions: Other: Grape
- Treatment (Experimental): Grape or Placebo
  Interventions: Other: Grape

INTERVENTIONS:
Other: Grape — Reconstituted whole grape powder

SUMMARY:
This study investigated the effects of time-of-day of grape consumption on high-fat meal-induced oxidative stress.

DETAILED DESCRIPTION:
Grape consumption acts on the immune system to produce antioxidant and anti-inflammatory effects. Since immune activity demonstrates circadian rhythmicity, with peak activity occurring during waking hours, the timing of grape intake may influence the magnitude of its antioxidant effect. This study followed a 2 x 2 factorial randomized, controlled design wherein healthy men and women (n = 32) consumed either a grape or placebo drink with a high-fat meal in the morning or evening. Urine was collected for measurements of biomarkers of oxidative stress and grape metabolites at baseline and post-meal at hour 1 and hours 1-6

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 18-50 y

Exclusion Criteria:

* Employed in shift or night work
* Extreme early or late chronotype
* Presence of acute infection or chronic inflammatory disease
* Smoking
* Heavy aerobic exerciser
* Greater than moderate alcohol intake
* Pregnancy or lactation
* Use of non-steroidal anti-inflammatory medications or antioxidant dietary supplements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Urine F2-isoprostane | baseline
  Oxidative stress marker
Urine F2-isoprostane | hour 1
  Oxidative stress marker
Urine F2-isoprostane | hours 1-6
  Oxidative stress marker

CONTACTS AND LOCATIONS:
Locations (1):
- Idaho State University, Pocatello, Idaho, United States

IPD SHARING:
Plan to Share IPD: No